CLINICAL TRIAL: NCT01860612
Title: Safety and Effectiveness of the CustomFlex Artificial Iris Prosthesis for the Treatment of Iris Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Consultants, Inc. (Industry)
Collaborators: HumanOptics AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-001
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Full Aniridia; Partial Aniridia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- PMA Cohort (Experimental): Study participants that meet the inclusion/exclusion criteria for the study may be enrolled in the compassionate use treatment arm. The artificial iris will be implanted in the eye with an iris defect. The fellow eye can be treated 1 month after the primary eye.
  Interventions: Device: Artificial Iris (CustomFlex)
- Compassionate Use Cohort (Experimental): Study participants that do not meet the inclusion/exclusion criteria for the study may be enrolled in the compassionate use treatment arm. The artificial iris will be implanted in the eye with an iris defect. The fellow eye can be treated 1 month after the primary eye.
  Interventions: Device: Artificial Iris (CustomFlex)
- Continued Access Cohort (Experimental): Study participants that meet the inclusion/exclusion criteria for the study may be enrolled in the Continued Access cohort, after enrollment in the PMA cohort is complete.The fellow eye can be treated 1 month after the primary eye.
  Interventions: Device: Artificial Iris (CustomFlex)

INTERVENTIONS:
Device: Artificial Iris (CustomFlex)

SUMMARY:
The purpose of this study is to study the long term safety and effectiveness of an artificial iris prosthesis for the treatment of iris defects.

ELIGIBILITY:
Inclusion Criteria:

For the IDE study, subjects in whom the subject and study eye meet all of the following criteria were candidates for the PMA cohort of this study, or the Continued Access cohort after the PMA cohort was enrolled:

1. 22 years of age or older
2. Having a diagnosis of congenital or acquired full or partial iris defect in the study eye.
3. Having symptoms of light sensitivity, photophobia, and/or glare in the study eye.
4. Subjects should be pseudophakic, aphakic or require cataract extraction.
5. Signed and received a copy of the signed written informed consent.
6. Willingness and ability to comply with schedule for follow-up visits and postoperative evaluations.

All adult and pediatric subjects who participated in the 12-month AI-001 IDE clinical trial who meet the following inclusion criteria are eligible for enrollment in the PAS; hereafter referred to as the "Long Term Extension Cohort":

1. Previous AI-001 IDE study participant who was enrolled before PMA approval (i.e., before May 30, 2018) and has had the CustomFlex™ Artificial Iris implanted for 36 months or less if enrolled as an adult or for 60 months or less if enrolled as a pediatric subject.
2. Signed and received a copy of the signed written informed consent.
3. Willingness and ability to comply with schedule for follow-up visits and postoperative evaluations.

Pediatric subjects in whom the subject and study eye meet all of the following criteria are candidates for enrollment in the Pediatric New Enrollment Cohort:

1. Age between 3 years and less than 22 years at the time of consent for the OSB PAS.
2. Having a diagnosis of congenital or acquired full or partial iris defect in the study eye.
3. Having symptoms of light sensitivity, photophobia, and/or glare or other aniridic symptoms in the study eye.
4. Subjects should be pseudophakic, aphakic or require cataract extraction.
5. Signed and received a copy of the signed written informed consent for the OSB PAS.
6. Willingness and ability to comply with schedule for follow-up visits and postoperative evaluations.

Exclusion Criteria:

There are no exclusion criteria for the Long Term Extension Cohort .

For the IDE study, all subjects in whom the subject or study eye meets any of the following criteria will were excluded from the PMA cohort of this study, or the Continued Access cohort after the PMA cohort was enrolled:

1. Uncontrolled ocular inflammation (e.g., uveitis).
2. Preoperative intraocular pressure > 21 mm Hg.
3. Subjects with a current condition that, in the investigator's opinion, would interfere with the treatment.
4. Subjects with any of the following conditions:

   1. Severe chronic uveitis
   2. Microphthalmus
   3. Untreated retinal detachment
   4. Untreated chronic glaucoma
   5. Rubella cataract
   6. Rubeosis of the iris
   7. Proliferative diabetic retinopathy
5. Female subjects who are pregnant or lactating at the time of surgery.
6. Subjects with a known sensitivity to required postoperative study medications (4th generation fluoroquinolone or steroid anti-inflammatory) if an alternative medication is not available.
7. Subjects under legal guardianship or who, in the investigator's opinion, lack the mental capacity to provide written informed consent for study participation.
8. Stargardt's retinopathy.
9. Subjects with gastric ulcers or diabetes mellitus in whom high doses of postoperative systemic steroids are required.
10. Surgical difficulty of the planned surgery, which might increase the potential for complications.
11. No useful vision or vision potential in the fellow eye.
12. Clear crystalline lens (in eyes with intact natural, crystalline lens).
13. Implantation of a CustomFlex™ Artificial Iris prosthesis in the contralateral eye within the previous 4 weeks.
14. In the investigator's opinion, the presence of a condition or finding in the contralateral eye that would make it unsafe to implant a CustomFlex™ Artificial Iris prosthesis in the study eye.

All pediatric subjects in whom the subject or study eye meets any of the following criteria will be excluded from enrollment in the Pediatric New Enrollment Cohort:

1. Uncontrolled ocular inflammation (e.g., uveitis).
2. Preoperative intraocular pressure > 21 mm Hg.
3. Subjects with a current condition that, in the investigator's opinion, would interfere with the treatment.
4. Subjects with any of the following conditions:

   1. Severe chronic uveitis
   2. Microphthalmus
   3. Untreated retinal detachment
   4. Untreated chronic glaucoma
   5. Rubella cataract
   6. Rubeosis of the iris
   7. Proliferative diabetic retinopathy
   8. Intraocular infections
5. Severe endothelial corneal dystrophy.
6. Subjects in whom an ocular surgery to treat an existing condition is planned to be performed in the study eye within 6 months after the artificial iris implant surgery day.
7. Female subjects who are pregnant or lactating at the time of surgery.
8. Subjects with a known sensitivity to required postoperative study medications (4th generation fluoroquinolone or steroid anti-inflammatory) if an alternative medication is not available.
9. Subjects under legal guardianship or who, in the investigator's opinion, lack the mental capacity to provide written informed consent for study participation.
10. Stargardt's retinopathy.
11. Subjects with gastric ulcers or diabetes mellitus in whom high doses of postoperative systemic steroids are required.
12. Surgical difficulty of the planned surgery, which might increase the potential for complications.
13. No useful vision or vision potential in the fellow eye.
14. Clear crystalline lens (in eyes with intact natural, crystalline lens).
15. Implantation of a CustomFlex™ Artificial Iris prosthesis in the contralateral eye within the previous 4 weeks.
16. In the investigator's opinion, the presence of a condition or finding in the contralateral eye that would make it unsafe to implant a CustomFlex™ Artificial Iris prosthesis in the study eye.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Symptoms | SCR & 6 Month
  Quality of vision will be assessed using the National Eye Institute Visual Functioning Questionnaire - 25.
Participant Satisfaction | SCR & 6 Month
  Participant satisfaction will be assessed using the Global Aesthetic Improvement Scale.
Complications and Adverse Events | SCR & 6 Month
  Complications and adverse events will be assessed through tabulation of adverse events, changes in vision, cell density, intraocular pressure, and slit lamp exam.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Advanced Vision Care, Los Angeles, California
  - Jules Stein Eye Institute, Los Angeles, California
  - Woolfson Eye Institute, Atlanta, Georgia
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - Price Vision Group, Indianapolis, Indiana
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - The Mackool Eye Institute, Astoria, New York
  - Rosenthal Eye Surgery, Great Neck, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Oregon Eye Associates, Eugene, Oregon
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - Alkek Eye Center/ Baylor College of Medicine, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah